CLINICAL TRIAL: NCT01699633
Title: Effect of Rifampin-containing Anti-TB Therapy on Nevirapine Plasma Pharmacokinetics in HIV/TB Co-infected Children < 3 Years Old
Brief Title: Rifampin and Nevirapine Interactions in Young Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PK-TBHIV02; R01HD071779 (NIH)
Record Dates: First submitted 2012-09-14; First posted 2012-10-04 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Tuberculosis; HIV
Keywords: Drug-drug interactions; Drug-gene interactions; Nevirapine; Rifampicin; children
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Plasma Whole blood DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Nevirapine is the preferred nonnucleoside reverse transcriptase inhibitor (NNRTI) for treatment of HIV in children younger than 3 years old who have tuberculosis (TB) coinfection. However, there is very limited data on the drug-drug interactions between rifampin and nevirapine in children of this age group. The purpose of this study is to determine the effect of rifampin-containing anti-TB treatment on the blood levels of nevirapine in young children with HIV and TB coinfection. Also, the study will find out whether checking the genetic makeup of a child could help to determine the appropriate dose of nevirapine in the setting of concomitant anti-TB treatment.

DETAILED DESCRIPTION:
HIV and TB coinfection is a common and a major cause of death in children globally. Treatment of the two infections together at the same time saves lives but some of the TB medications have significant drug-drug interactions with commonly used antiretroviral drugs (ARVs). Rifampin induces the activity of cytochorme P450 (CYP) enzymes and may reduce the blood levels of important ARVs such as nevirapine or efavirenz when coadministered. The CYP enzymes activity can vary from person to person depending on genetic makeup, further complicating drug-drug interactions. Nevirapine undergoes extensive metabolism by hepatic CYP3A and CYP2B6 enzymes. The induction of CYP3A4 and 2B6 by rifampin causes a 10 - 68% reduction in nevirapine exposure upon concomitant dosing in adults. Pharmacokinetic studies suggest that nevirapine trough concentrations in HIV-infected children tend to be lower or sub-therapeutic in children younger than 3 years old. To our knowledge, the only study that evaluated the influence of rifampin on nevirapine plasma concentrations in younger children reported substantial reductions in nevirapine concentrations with rifampin co-administration. It is currently unclear whether using the recommended nevirapine dose (200 mg/m2 twice daily) without the two-week lead-in of 200 mg/m2 once daily will overcome the risk of sub-therapeutic concentrations in the setting of concomitant anti-TB treatment. This study will investigate the effect of rifampin-containing anti-TB therapy on nevirapine plasma concentration in children younger than 3 years old, as well as find out whether CYP2B6 and CYP3A4 enzymes genetic polymorphisms influence the magnitude of the drug-drug interactions.

Specific hypotheses to be tested are:

1. Rifampin-containing anti-TB therapy substantially reduces nevirapine Cmin and estimated AUC0-12h in young HIV-infected children (by at least 40%).
2. CYP2B6 extensive metabolizers have substantially lower plasma nevirapine Cmin and estimated AUC0-12h in the presence than in the absence of rifampin-containing TB therapy, but no significant difference in intermediate and slow metabolizers.

A two-arm parallel assignment pharmacokinetic study in TB/HIV co-infected children will be performed at the KATH. Children aged 3 - 35 months with HIV infection with or without TB coinfection, antiretroviral therapy (ART)-naïve, not previously exposed to nevirapine will be enrolled. The ART regimen will consist of nevirapine 200 mg/m2 plus zidovudine (ZDV) 180 - 240 mg/m2 and lamivudine (3TC) 4 mg/kg twice daily in accordance with WHO guidelines. There will be no lead-in dosing of nevirapine in the co-infected patients on rifampin. The dose of nevirapine in the HIV mono-infected group will be 200 mg/m2 daily x 2 weeks and then twice daily afterwards. Standard anti-TB therapy will be prescribed to the HIV/TB co-infected patients. Anti-TB treatment will start immediately upon diagnosis. Antiretroviral therapy will be started as soon as anti-TB therapy is tolerated (typically within 2 to 8 weeks).

A complete medical history, physical examination, and staging of HIV disease will be performed before initiation of ART and at subsequent study visits. Relevant data will be collected using standardized forms. Baseline measurements prior to initiation of ART will include complete blood count (CBC), blood urea nitrogen, creatinine, liver function tests (LFTs), CD4 cell count determination and plasma HIV-1 RNA level. Measurements of CD4 cell count and plasma HIV-1 RNA will be repeated at weeks 12 and 24 after starting ART. All study participants will follow-up at 2 and 4 weeks, as well as monthly for assessment of treatment side effects. Additional tests will be done when clinically indicated to evaluate for drug toxicity.

Pharmacokinetic testing will be performed at week 4 of ART in both arms and at 4 weeks after anti-TB treatment is stopped while the child is receiving ART only in the HIV/TB co-infected group. All patients will be admitted to the hospital the night prior to complete PK sampling. Study drugs will be administered after at least a 2-hour fast in non-breastfed children. Younger children on exclusive breast-feeding will be allowed to breast feed as needed throughout the study. At each sampling time, 2 mL of blood will be collected into an EDTA tube at times 0, 2, 6 and 12 hours post-dose for determination of nevirapine concentrations. Actual times of sampling will be recorded. The blood samples will be centrifuged at 3000g for 10 minutes and plasma stored at - 70oC until measurement of plasma drug concentrations. Nevirapine concentrations in plasma will be measured using validated gas chromatography with mass spectrometry and nonlinear mixed-effects modeling (using NONMEM, version VI) will be used to estimate pharmacokinetic parameters (CL/F, AUC, Cmin, Cmax), inter-individual error, and residual error. DNA sample will stored for genotyping of drug metabolizing enzymes and transporters.

ELIGIBILITY:
Inclusion Criteria:

1. HIV seropositive children with or without active TB
2. Aged 3 to 35 months old
3. Antiretroviral-naïve and meet criteria for initiation of antiretroviral therapy
4. Are available for follow-up until achievement of a study endpoint like completion of study or discontinuation of HAART, and/or PK sampling

Exclusion Criteria:

1. Unable to obtain informed signed consent parent(s) or legal guardian
2. Have AIDS-related opportunistic infections other than TB, history of or proven acute hepatitis within 30 days of study entry, persistent vomiting, or diarrhea
3. Hemoglobin < 6 g/dl, white blood cells < 2500/mm3, serum creatinine > 1.5 mg/dl, AST and ALT > 2X upper limit of normal.

Ages: 3 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3 to 35 months with HIV infection with or without TB
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Area under time curve (AUC) of nevirapine | At week of 4 of HIV therapy
  Compare nevirapine AUC0-12h between HIV-infected children without TB and those with TB, as well as in the absence of and presence of rifampin-containing anti-TB therapy in co-infected patients

SECONDARY OUTCOMES:
Number of children with grade 3 or 4 liver enzymes elevations compared to baseline, new onset of skin rash, nausea, vomiting or treatment modification due to drug side effects | Up to week 24 of HIV therapy
  Compare frequency of adverse events as a measure of safety and tolerability between HIV-infected children with and without TB coinfection
Number of children with nevirapine 12-hour post-dose concentration (C12h) < 3000 ng/mL | Week 4 of HIV therapy
  Relationship between clinical factors (weight, gender, nutritional status) as well as genetic factors (CYP2B6, CYP3A4 polymorphisms) and nevirapine C12h will be investigated
Time to HIV-1 RNA suppression below 50 copies/mL and change in CD4 cell count from baseline | Up to week 24 of HIV therapy
  Relationship between nevirapine pharmacokinetics (AUC0-12h, C12h) and time to virologic suppression as well as increase in CD4 cell count from baseline in the combined study population
Peak concentration (Cmax) and concentration at 12-hours (C12h) post-dose of nevirapine | At week 4 of therapy
  Compare nevirapine Cmax and C12h between HIV-infected children without TB and those with TB, as well as in the absence of and presence of rifampin-containing anti-TB therapy in co-infected patients

CONTACTS AND LOCATIONS:
Overall Officials: Awewura Kwara, MD, MPH&TM, Principal Investigator — The Miriam Hospital
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ghana

REFERENCES:
- [Derived] Enimil A, Antwi S, Yang H, Dompreh A, Alghamdi WA, Gillani FS, Orstin A, Bosomtwe D, Opoku T, Norman J, Wiesner L, Langaee T, Peloquin CA, Court MH, Greenblatt DJ, Kwara A. Effect of First-Line Antituberculosis Therapy on Nevirapine Pharmacokinetics in Children Younger than Three Years Old. Antimicrob Agents Chemother. 2019 Sep 23;63(10):e00839-19. doi: 10.1128/AAC.00839-19. Print 2019 Oct. PMID 31332062